CLINICAL TRIAL: NCT01946165
Title: A Pre-Operative Study to Assess the Effects of Abiraterone Acetate Plus LHRH Agonist and Abiraterone Acetate Plus LHRH Agonist and Enzalutamide for Six Months for Prostate Cancer Patients at High-Risk for Recurrence
Brief Title: Abiraterone Acetate Plus LHRH Agonist and Abiraterone Acetate Plus LHRH Agonist and Enzalutamide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Janssen Services, LLC (Industry); Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0332; NCI-2014-01041 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Results first posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; High risk prostate cancer; Abiraterone acetate; Zytiga; Prednisone; Enzalutamide; MDV3100; XTANDI; Androgen ablation; LHRHa; Hormonal therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abiraterone Acetate + Prednisone + Enzalutamide + LHRHa (Experimental): Patients receive abiraterone acetate (1,000 mg daily) plus prednisone (5mg once daily) in combination with enzalutamide (160 mg daily) and LHRHa. Patients receive a LHRHa (monthly injection or three-month injection) for a maximum of 7 months before a prostatectomy is performed. Study doctor will decide what hormone therapy patient receives.
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone; Drug: Enzalutamide; Drug: LHRHa
- Abiraterone Acetate + Prednisone + LHRHa (Experimental): Patients receive abiraterone acetate (1,000 mg daily) plus prednisone (5mg once daily) and LHRHa. Patients receive a LHRHa (monthly injection or three-month injection) for a maximum of 7 months before a prostatectomy is performed. Study doctor will decide what hormone therapy patient receives.
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone; Drug: LHRHa

INTERVENTIONS:
Drug: Abiraterone Acetate — 1,000 mg by mouth daily for each 28 day cycle.
  Other Names: Zytiga
Drug: Prednisone — 5 mg by mouth once daily for each 28 day cycle.
Drug: Enzalutamide — 160 mg by mouth daily for each 28 day cycle.
  Other Names: MDV3100; XTANDI
  Arms: Abiraterone Acetate + Prednisone + Enzalutamide + LHRHa
Drug: LHRHa — Patients receive a LHRHa (monthly injection or three-month injection) for a maximum of 7 months before a prostatectomy is performed. Study doctor will decide what hormone therapy patient receives.

SUMMARY:
The goal of this clinical research study is to learn if adding the combination of abiraterone acetate and prednisone with or without enzalutamide to hormonal therapy can help to control prostate cancer when given before surgery. The safety of the drug combination will also be studied.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (like the roll of dice) to 1 of 2 groups. You will have a 2 out of 3 chance of being assigned to Group A and a 1 out of 3 chance of being assigned to Group B.

If you are in Group A, you will receive hormonal therapy (LHRH), abiraterone acetate, prednisone, and enzalutamide.

If you are in Group B, you will receive LHRH, abiraterone acetate, and prednisone.

Study Drug Administration:

The study doctor will decide what hormone therapy you will receive, will explain when and how you should take it, and explain any risks.

In addition, you will take 4 abiraterone acetate tablets by mouth each day (all at the same time) at least 1 hour before a meal or 2 hours after a meal. You will also take 1 tablet of prednisone by mouth 1 time each day to help lower the risk of side effects caused by abiraterone acetate.

If you are in Group A, you will also take 4 capsules of enzalutamide by mouth each day. You should take enzalutamide at about the same time every morning. Enzalutamide can be taken with or without food. If you miss a dose, you should NOT take another dose until the next day. You should tell the study doctor as soon as possible if you miss a dose.

About every 28-days is called a cycle. You should return all unused study drug and/or empty pill bottles at the end of each cycle.

Study Visits:

On Day 1 of Cycle 1:

* You will have a physical exam.
* Blood (about 3-4 tablespoons) will be drawn for routine tests and to check your prostatic specific antigen (PSA) level.

On Day 15 of Cycles 1, 2 and 3, blood (about 2 tablespoons) will be drawn to check your liver function. These tests may be done at your local doctor's office and the results faxed to MD Anderson.

On Day 1 of Cycles 2, 3, 4, 5 and 6:

* You will have a physical exam.
* Blood (about 3-4 tablespoons) will be drawn for routine tests. This blood will also be used to check your PSA level.

The testing on Cycles 2, 4 and 6 may be done at your local doctor's office and the results faxed to MD Anderson.

Within 14 days before surgery and at your End of Treatment Visit:

* You will have a physical exam.
* Blood (about 3-4 tablespoons) and urine will be collected for routine tests. This blood will also be used to check your PSA level, your blood sugar levels, and blood-clotting function. You will be asked to fast for at least 8 hours before these blood draws.
* You will have a chest x-ray or a CT scan of the chest.
* You will have an EKG to check your heart function.

Surgery:

After 6 cycles of study treatment, you will have surgery to remove your prostate. You will be asked to sign a separate consent form for this surgery, and the risks will be discussed with you. Your leftover prostate gland tissue from surgery will be collected and used for biomarker testing.

About 4 to 8 weeks after your surgery:

* You will have a physical exam.
* Blood (about 3-4 tablespoons) drawn for routine tests. This blood will also be used to check your PSA, testosterone, cholesterol, and blood sugar levels.

Length of Study:

You may receive the study drugs for about 6 months. You will be taken off study early if the disease gets worse, if you have intolerable side effects, or if your study doctor thinks it is in your best interest to stop, or of you are unable to follow study directions.

Your participation on the study will be over once you have completed the visits after surgery.

This is an investigational study. Abiraterone acetate is FDA approved in combination with prednisone for the treatment of patients with metastatic castration-resistant prostate cancer who have received prior chemotherapy containing docetaxel. Prednisone is FDA approved and commercially available as a corticosteroid. Enzalutamide is FDA approved and commercially available for the treatment of certain types of prostate cancer. Their combination with hormone therapy in patients with prostate cancer is investigational.

Up to 69 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing/able to adhere to the prohibitions and restrictions specified in this protocol
2. Have signed an informed consent document indicating that the subjects understand the purpose of and procedures required for the study and are willing to participate in the study
3. Written Authorization for Use and Release of Health and Research Study Information has been obtained.
4. Male age >/=18 years.
5. Histologically or cytologically confirmed adenocarcinoma of the prostate with no histological variants (such as small cell, sarcomatoid, pure ductal cancer, transitional cell carcinoma).
6. Pathology review at treating academic institution or member institution (Note: if patient's prostate biopsy was not read at the treating institution, it must be reviewed at the study site to confirm eligibility).
7. At least three core biopsies involved with cancer (a minimum of 6 core biopsies must be obtained at baseline). A prostate biopsy within 3 months from screening is allowed for entry requirements. Patients must have a Gleason score > 5 (total).
8. At least one of the following features: a) PSA > 10 ng/ml; b) PSA velocity > 2 ng/ml/year (defined as a rise in PSA of > 2 ng/ml in the preceding 12 month period); c) Gleason score >/= 7; d) Gleason score 6 if either PSA >/= 10 ng/ml or PSA velocity >/=2 ng/ml/year
9. Serum testosterone >200 ng/dL. For patients treated with up to 1 month of LHRH agonist, a testosterone measurement prior to the LHRH treatment will be used to determine eligibility, and must have been > 200 ng/dL.
10. Urologist must agree that patient is suitable for prostatectomy.
11. No evidence of metastatic disease as determined by imaging procedures.
12. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
13. Hemoglobin >/= 10.0 g/dL independent of transfusion.
14. Platelet count >/=100,000/µL.
15. Patients should have adequate bone marrow function defined as an absolute peripheral neutrophil count (ANC) >/= 1,500.
16. Creatinine clearance >/= 60 mL/min
17. Serum potassium >/= 3.5 mmol/L.
18. Serum albumin >/= 3.5 g/dL.
19. Liver function test with serum bilirubin </= 1.5x upper limit of normal (ULN) and ALT and AST </= 1.5x ULN.
20. Able to swallow the study drug whole as a tablet.
21. Patients must have normal coagulation profile and no history of substantial non- iatrogenic bleeding diathesis.
22. Agree to use a double-barrier method of contraception which involves the use of a condom in combination with one of the following: contraceptive sponge, diaphragm, or cervical ring with spermicidal gel or foam, if having sex with a woman of child-bearing potential during the length of the study and for one week after abiraterone is discontinued and for at least three months after enzalutamide is discontinued.
23. Willing to take abiraterone acetate on an empty stomach; no food should be consumed at least two hours before and for at least one hour after the dose of abiraterone acetate is taken.

Exclusion Criteria:

1. Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection.
2. Chronically uncontrolled hypertension, defined conventionally as consistent systolic pressures above 140 or diastolic pressures above 90 despite anti-hypertensive therapy. Note that this is NOT a criterion related to particular BP results at the time of assessment for eligibility, nor does it apply to acute BP excursions that are related to iatrogenic causes, acute pain or other transient, reversible causes.
3. Requirement for corticosteroids greater than the equivalent of 5 mg of prednisone daily.
4. Poorly controlled diabetes defined by Hemoglobin A1C > 7.0 at screening.
5. Active or symptomatic viral hepatitis or chronic liver disease.
6. History of pituitary or adrenal dysfunction.
7. Clinically significant cardiovascular disease including: a) Myocardial infarction within 6 months of Screening visit; b) Uncontrolled angina within 3 months of Screening visit; c) Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or subjects with history of congestive heart failure NYHA class 3 or 4 in the past, or history of anthracycline or anthracenedione (mitoxantrone) treatment, unless a screening echocardiogram or multi-gated acquisition scan (MUGA) performed within three months of the Screening visit results in a left ventricular ejection fraction that is >/= 50%; d) History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsade de pointes); e) Prolonged corrected QT interval by the Fridericia correction formula (QTcF) on the screening Electrocardiogram (ECG) > 470 msec; f) History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place;
8. (Exclusion #7 continued): g) Hypotension (systolic blood pressure < 86 mmHg or bradycardia with a heart rate of <50 beats per minute on the Screening ECG, unless pharmaceutically induced and thus reversible (i.e. beta blockers).
9. Other malignancy, except non-melanoma skin cancer, that is active or has a >/= 30% probability of recurrence within 12 months.
10. History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug.
11. Prior hormone therapy for prostate cancer including orchiectomy, antiandrogens, ketoconazole, or estrogens (5-alpha reductase inhibitors allowed), or LHRH agonists/antagonists (*Note: LHRH allowed if begun within 1 month of Day 1). Patients having previous or current antiandrogen treatment of greater than 4 weeks in duration prior to Cycle 1 Day 1 are eligible with appropriate washout.
12. Prior systemic treatment with an azole drug within four weeks of Cycle 1 Day1.
13. Current enrollment in an investigational drug or device study or participation in such a study within 30 days of Cycle 1 Day 1.
14. Allergies, hypersensitivity, or intolerance to prednisone, LHRH analog or excipients of prednisone LHRH analog, and abiraterone acetate and enzalutamide.
15. Previous use of abiraterone acetate or other investigational CYP17 inhibitor (e.g., TAK-700).
16. Previous investigational antiandrogens (e.g., Enzalutamide, BMS-641988).
17. Patients receiving anti-coagulant therapy who are unable to stop prior to surgery.
18. Condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with patient's participation in the study.
19. Severely compromised immunological state, including being positive for the human immunodeficiency virus (HIV).
20. Patients who are not appropriate surgical candidates for radical prostatectomy based on the evaluation of co-existent medical diseases and competing potential causes of death (such as but not limited to, unstable angina, myocardial infarction within the previous 6 months, or use of ongoing maintenance therapy for life-threatening ventricular arrhythmia, uncontrolled hypertension).
21. Prior chemotherapy, radiation or immune therapy for prostate cancer.
22. Patients unable to tolerate transrectal ultrasound.
23. Concomitant therapy with any of the following: a) Chemotherapeutic, biologic, or other agents with anti-tumor activity against prostate cancer other than assigned study drug; b) Anti-androgens (steroidal or non-steroidal) such as cyproterone acetate, flutamide, nilutamide, bicalutamide, etc. other than assigned study drug; c) 5-alpha reductase inhibitors such as finasteride, dutasteride, anabolic steroids, etc.; d) Estrogens, progestational agents such as megestrol, medroxyprogesterone, DES, cyproterone, spironolactone > 50 mg/kg, etc.; e) Androgens such as testosterone, dehydroepiandrosterone [DHEA], etc.; f) Ketoconazole; g) Herbal products that may decrease PSA levels (e.g., saw palmetto)
24. Active infection or other medical condition that would make prednisone/ prednisolone (corticosteroid) use contraindicated.
25. Severe hepatic impairment (Child-Pugh Class C).
26. History of seizure or any condition that may predispose to seizure including, but not limited to underlying brain injury, stroke, primary brain tumors, brain metastases, or alcoholism. Also, history of loss of consciousness or transient ischemic attack within 12 months of enrollment (Day 1 visit).
27. History of significant bleeding disorder unrelated to cancer, including: a) Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease); b) Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies) of Screening visit; c) History of GI bleeding within 6 months of Screening visit.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Logothetis, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Han H, Wang Y, Curto J, Gurrapu S, Laudato S, Rumandla A, Chakraborty G, Wang X, Chen H, Jiang Y, Kumar D, Caggiano EG, Capogiri M, Zhang B, Ji Y, Maity SN, Hu M, Bai S, Aparicio AM, Efstathiou E, Logothetis CJ, Navin N, Navone NM, Chen Y, Giancotti FG. Mesenchymal and stem-like prostate cancer linked to therapy-induced lineage plasticity and metastasis. Cell Rep. 2022 Apr 5;39(1):110595. doi: 10.1016/j.celrep.2022.110595. PMID 35385726
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with prostate cancer at high-risk for recurrence randomized to two treatment groups
Pre-assignment Details: Out of 69 participants, due to a screen failure, no arm assignment was made for 1 participant; therefore, only 68 participants were treated and evaluable for outcome analysis.
Groups:
- Group A: Abiraterone + Enzalutamide + LHRHa + Prednisone.: Patients receive abiraterone acetate (1,000 mg daily) plus prednisone (5mg once daily) and LHRHa. Patients receive a LHRHa (monthly injection or three-month injection) for a maximum of 7 months before a prostatectomy is performed. Study doctor will decide what hormone therapy patient receives.
  Abiraterone Acetate: 1,000 mg by mouth daily for each 28 day cycle.
  Prednisone: 5 mg by mouth once daily for each 28 day cycle.
  Enzalutamide: 160 mg by mouth daily for each 28 day cycle.
  LHRHa: Patients receive a LHRHa (monthly injection or three-month injection) for a maximum of 7 months before a prostatectomy is performed. Study doctor will decide what hormone therapy patient receives.
- Group B: Abiraterone + LHRHa + Prednisone.: Patients receive abiraterone acetate (1,000 mg daily) plus prednisone (5mg once daily) and LHRHa. Patients receive a LHRHa (monthly injection or three-month injection) for a maximum of 7 months before a prostatectomy is performed. Study doctor will decide what hormone therapy patient receives.
  Abiraterone Acetate: 1,000 mg by mouth daily for each 28 day cycle.
  Prednisone: 5 mg by mouth once daily for each 28 day cycle.
  LHRHa: Patients receive a LHRHa (monthly injection or three-month injection) for a maximum of 7 months before a prostatectomy is performed. Study doctor will decide what hormone therapy patient receives.
Period: Overall Study
Arm/Group | Group A: Abiraterone + Enzalutamide + LHRHa + Prednisone. | Group B: Abiraterone + LHRHa + Prednisone.
Started | 45 | 23
Completed | 43 | 21
Not Completed | 2 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group A: Abiraterone + Enzalutamide+ LHRHa+ Prednisone: Patients receive abiraterone acetate (1,000 mg daily) plus prednisone (5mg once daily) in combination with enzalutamide (160 mg daily) and LHRHa. Patients receive a LHRHa (monthly injection or three-month injection) for a maximum of 7 months before a prostatectomy is performed. Study doctor will decide what hormone therapy patient receives.
  Abiraterone Acetate: 1,000 mg by mouth daily for each 28 day cycle.
  Prednisone: 5 mg by mouth once daily for each 28 day cycle.
  Enzalutamide: 160 mg by mouth daily for each 28 day cycle.
  LHRHa: Patients receive a LHRHa (monthly injection or three-month injection) for a maximum of 7 months before a prostatectomy is performed. Study doctor will decide what hormone therapy patient receives.
- Group B: Abiraterone+ LHRHa+ Prednisone: Patients receive abiraterone acetate (1,000 mg daily) plus prednisone (5mg once daily) and LHRHa. Patients receive a LHRHa (monthly injection or three-month injection) for a maximum of 7 months before a prostatectomy is performed. Study doctor will decide what hormone therapy patient receives.
  Abiraterone Acetate: 1,000 mg by mouth daily for each 28 day cycle.
  Prednisone: 5 mg by mouth once daily for each 28 day cycle.
  LHRHa: Patients receive a LHRHa (monthly injection or three-month injection) for a maximum of 7 months before a prostatectomy is performed. Study doctor will decide what hormone therapy patient receives.
- Total: Total of all reporting groups
Arm/Group | Group A: Abiraterone + Enzalutamide+ LHRHa+ Prednisone | Group B: Abiraterone+ LHRHa+ Prednisone | Total
Number analyzed (Participants) | 45 | 23 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 12 | 36
  >=65 years | 21 | 11 | 32
Age, Continuous [Median (Full Range); unit: years] | 66 [47 to 75] | 64 [49 to 74] | 65 [47 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 45 | 23 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 32 | 16 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 45 | 23 | 68

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Pathologic Stage Less Than or Equal to ypT2N0
Description: The proportion of participants with pathologic stage less than or equal to ypT2N0 will be descriptively summarized and compared between the two treatment arms. The proportion will be calculated as the number of patients with less than or equal to ypT2N0 in each treatment arm divided by the total number of patients who underwent surgery in the same arm.
Time Frame: For all participants who underwent surgery, from start of treatment until surgery is completed
Population: Patients that are evaluable are included in these values.
Measure: Count of Participants; unit: Participants
Groups:
- Group A: Abiraterone + Enzalutamide + LHRHa + Prednisone.: Patients receive abiraterone acetate (1,000 mg daily) plus prednisone (5mg once daily) in combination with enzalutamide (160 mg daily) and LHRHa. Patients receive a LHRHa (monthly injection or three-month injection) for a maximum of 7 months before a prostatectomy is performed. Study doctor will decide what hormone therapy patient receives.
  Abiraterone Acetate: 1,000 mg by mouth daily for each 28 day cycle.
  Prednisone: 5 mg by mouth once daily for each 28 day cycle.
  Enzalutamide: 160 mg by mouth daily for each 28 day cycle.
  LHRHa: Patients receive a LHRHa (monthly injection or three-month injection) for a maximum of 7 months before a prostatectomy is performed. Study doctor will decide what hormone therapy patient receives.
Arm/Group | Group A: Abiraterone + Enzalutamide + LHRHa + Prednisone. | Group B: Abiraterone + LHRHa + Prednisone
Number analyzed (Participants) | 43 | 21
Participants | 13 | 11

2. Secondary Outcome: Proportion of Participants With Positive Surgical Margins
Description: The difference in the rate of positive surgical margins between the two groups will be descriptively summarized.
Time Frame: For both groups, tumor samples collected at baseline and during surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Abiraterone + Enzalutamide + LHRHa + Prednisone | Group B: Abiraterone + LHRHa + Prednisone
Number analyzed (Participants) | 43 | 21
Participants | 9 | 2

ADVERSE EVENTS:
Time Frame: From informed consent to 4 weeks after the patient has stopped treatment
Description: Adverse events were collected and reported according to protocol requirements.
Groups:
- Arm A: Abiraterone + Enzalutamide + LHRHa + Prednisone: Patients receive abiraterone acetate (1,000 mg daily) plus prednisone (5mg once daily) in combination with enzalutamide (160 mg daily) and LHRHa. Patients receive a LHRHa (monthly injection or three-month injection) for a maximum of 7 months before a prostatectomy is performed. Study doctor will decide what hormone therapy patient receives.
  Abiraterone Acetate: 1,000 mg by mouth daily for each 28 day cycle.
  Prednisone: 5 mg by mouth once daily for each 28 day cycle.
  Enzalutamide: 160 mg by mouth daily for each 28 day cycle.
  LHRHa: Patients receive a LHRHa (monthly injection or three-month injection) for a maximum of 7 months before a prostatectomy is performed. Study doctor will decide what hormone therapy patient receives.
Arm/Group | Arm A: Abiraterone + Enzalutamide + LHRHa + Prednisone | Group B: Abiraterone + LHRHa + Prednisone
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/23
Serious Adverse Events (participants affected / at risk) | 4/45 | 1/23
Other Adverse Events (participants affected / at risk) | 45/45 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Abiraterone + Enzalutamide + LHRHa + Prednisone (N=45) | Group B: Abiraterone + LHRHa + Prednisone (N=23)
pancreatitis (Metabolism and nutrition disorders) | 1 | 0
possible mini stroke (Cardiac disorders) | 1 | 0
PE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
abdominal pain (Vascular disorders) | 1 | 0
neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
hematoma (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Abiraterone + Enzalutamide + LHRHa + Prednisone (N=45) | Group B: Abiraterone + LHRHa + Prednisone (N=23)
Abdominal pain (Vascular disorders) | 3 | 3
Agitation (Psychiatric disorders) | 1 | 1
Alanine aminotransferase increased (Hepatobiliary disorders) | 37 | 12
Alkaline phosphatase increased (Investigations) | 5 | 1
Allergic reaction (Immune system disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 20 | 9
Anxiety (Psychiatric disorders) | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Aspartate aminotransferase increased (Hepatobiliary disorders) | 24 | 12
Atrial fibrillation (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bladder spasm (Renal and urinary disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 1
Blood bilirubin increased (Hepatobiliary disorders) | 10 | 10
Blurred vision (Eye disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 1
Cholesterol high (Investigations) | 7 | 5
Cognitive disturbance (Psychiatric disorders) | 4 | 0
Concentration impairment (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Creatinine increased (Investigations) | 1 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1
Depressed level of consciousness (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 5
Dizziness (Nervous system disorders) | 9 | 0
Dry eye (Eye disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Edema limbs (General disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 6 | 3
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Fatigue (General disorders) | 34 | 10
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1
Gait disturbance (General disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Hallucinations (Psychiatric disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 3
Hemoglobin (Blood and lymphatic system disorders) | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 0
Hot flashes (Vascular disorders) | 36 | 16
Hypercalcemia (Metabolism and nutrition disorders) | 8 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 30 | 15
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 2
Hypernatremia (Metabolism and nutrition disorders) | 12 | 8
Hypertension (Vascular disorders) | 14 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 10 | 3
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 12 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 12 | 4
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 5 | 1
Investigations - Other, specify (Investigations) | 4 | 0
Irritability (General disorders) | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 1
Lymphedema (Vascular disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 8 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 7 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 7 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 2 | 0
Platelet count decreased (Blood and lymphatic system disorders) | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Prostate infection (Infections and infestations) | 0 | 1
Proteinuria (Renal and urinary disorders) | 5 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 0
Psychosis (Psychiatric disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 1
Renal calculi (Renal and urinary disorders) | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 1
Scrotal pain (Reproductive system and breast disorders) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 1
Testicular pain (Reproductive system and breast disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Transient ischemic attacks (Nervous system disorders) | 1 | 0
Upper respiratory infection (Injury, poisoning and procedural complications) | 1 | 1
Urinary frequency (Renal and urinary disorders) | 16 | 7
Urinary incontinence (Renal and urinary disorders) | 10 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 3 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Watering eyes (Eye disorders) | 1 | 0
Weight loss (Metabolism and nutrition disorders) | 1 | 0
White blood cell decreased (Blood and lymphatic system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT01946165/Prot_SAP_000.pdf